CLINICAL TRIAL: NCT07293351
Title: ROSETTA RCC-208: A Phase 1/2 Open-label, Multi-center, Randomized Study of Pumitamig Alone or in Combination With Ipilimumab or Cabozantinib in Participants With Advanced Renal Cell Carcinoma (RCC)
Brief Title: A Study to Evaluate the Safety, Tolerability, and Efficacy of Pumitamig Alone or in Combination With Ipilimumab or Cabozantinib in Participants With Advanced Renal Cell Carcinoma (RCC) (ROSETTA RCC-208)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA266-0008; 2025-523637-26 (Other: EU CT Number); U1111-1327-6332 (Other: UTN)
Record Dates: First submitted 2025-12-17; First posted 2025-12-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Advanced Renal Cell Carcinoma (RCC)
Keywords: Renal Cell Carcinoma; Cabozantinib; Pumitamig; Ipilmumab; Nivolumab
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Ipilimumab; cabozantinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Part 1A: Arm A (Experimental)
  Interventions: Drug: Pumitamig; Drug: Ipilimumab
- Part 1A: Arm B (Experimental)
  Interventions: Drug: Pumitamig; Drug: Ipilimumab
- Part 1B: Arm G (Experimental)
  Interventions: Drug: Pumitamig; Drug: Cabozantinib
- Part 1B: Arm H (Experimental)
  Interventions: Drug: Pumitamig; Drug: Cabozantinib
- Part 2A: Arm C (Experimental)
  Interventions: Drug: Pumitamig; Drug: Ipilimumab
- Part 2A: Arm D (Experimental)
  Interventions: Drug: Pumitamig; Drug: Ipilimumab
- Part 2A: Arm E (Other)
  Interventions: Drug: Ipilimumab; Drug: Nivolumab
- Part 2A: Arm F (Experimental)
  Interventions: Drug: Pumitamig
- Part 2B: Arm I (Experimental)
  Interventions: Drug: Pumitamig; Drug: Cabozantinib
- Part 2B: Arm J (Experimental)
  Interventions: Drug: Pumitamig; Drug: Cabozantinib
- Part 2B: Arm K (Other)
  Interventions: Drug: Nivolumab
- Part 2B: Arm L (Experimental)
  Interventions: Drug: Pumitamig

INTERVENTIONS:
Drug: Pumitamig — Specified dose on specified days
  Other Names: BMS-986545
  Arms: Part 1A: Arm A; Part 1A: Arm B; Part 1B: Arm G; Part 1B: Arm H; Part 2A: Arm C; Part 2A: Arm D; Part 2A: Arm F; Part 2B: Arm I; Part 2B: Arm J; Part 2B: Arm L
Drug: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy
  Arms: Part 1A: Arm A; Part 1A: Arm B; Part 2A: Arm C; Part 2A: Arm D; Part 2A: Arm E
Drug: Cabozantinib — Specified dose on specified days
  Arms: Part 1B: Arm G; Part 1B: Arm H; Part 2B: Arm I; Part 2B: Arm J
Drug: Nivolumab — Specified dose on specified days
  Other Names: Opdivo
  Arms: Part 2A: Arm E; Part 2B: Arm K

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of Pumitamig alone or in combination with Ipilimumab or Cabozantinib in participants with advanced Renal Cell Carcinoma (RCC)

ELIGIBILITY:
Inclusion Criteria

* Participants must have a histologically confirmed diagnosis of locally advanced, unresectable (not amenable to curative surgery or radiation therapy) or metastatic Renal Cell Carcinoma (RCC).
* Participants must have clear cell RCC (ccRCC) or non-clear cell RCC (nccRCC) may be enrolled in Part 1. Note: Part 2 may only enroll participants with ccRCC.
* Participants may have favorable, intermediate or poor risk disease categories.
* Participants must not have received prior systemic therapy for metastatic RCC, with the following exceptions:

  i) One prior adjuvant or neoadjuvant therapy for completely resectable RCC is allowed if such therapy did not include an agent that targets vascular endothelial growth factor (VEGF) or VEGF receptors and if recurrence occurred at least 6 months after the last dose of adjuvant or neoadjuvant therapy.

ii) For Part 1A participants: Prior systemic therapy in the metastatic setting is allowed if the participant has not received any therapy targeting cytotoxic T-lymphocyte antigen 4 (CTLA-4) (e.g., ipilimumab).

iii) For Part 1B participants: Prior systemic therapy in the metastatic setting is allowed if the participant has not received prior treatment with cabozantinib.

- Participants must have measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

Exclusion Criteria

* Participants must not have any untreated known CNS metastases.
* Participants must not have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of Cycle 1 Day1 (C1D1).
* Participants must not have a history of interstitial lung disease or pneumonitis.
* Participants must not have an uncontrolled pleural or pericardial effusion requiring recurrent therapeutic drainage procedures.
* Participants must not have significant cardiovascular disease, such as myocardial infarction, unstable angina, arterial thrombosis, cerebrovascular accident within 6 months prior to C1D1, uncontrolled hypertension (≥ 150 systolic, ≥ 90 diastolic mm Hg) despite optimal medical management, or congenital long QT syndrome.
* Participants must not have a urine protein ≥ 2+ and 24 hour urine protein ≥ 1 g at baseline.
* Participants must not have evidence of major coagulation disorders.
* Participants must not have a history of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism within 6 months prior to C1D1.
* Participants must not have a history of abdominal fistula or gastrointestinal (GI) perforation within 6 months.
* Participants must not have had a major surgery or trauma within 28 days prior to C1D1.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2026-03-26 (Estimated); Primary Completion 2029-11-28 (Estimated); Study Completion 2031-11-26 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to approximately 2 years from end of treatment
  Phase 1
Number of participants with serious adverse events (SAEs) (as per Common Terminology Criteria for Adverse Events v5 (CTCAE v5)) | Up to approximately 2 years from end of treatment
  Phase 1
Number of participants with AEs meeting protocol-defined dose-limiting toxicity (DLT) criteria | Up to day 21 from first dose
  Phase 1
Number of participants with AEs leading to discontinuation | Up to approximately 2 years from end of treatment
  Phase 1
Number of participants with AEs leading to death | Up to approximately 2 years from end of treatment
  Phase 1
Objective response rate (ORR) (confirmed complete response (CR) or partial response (PR)) by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 per investigator assessment | Up to approximately 2 years from end of treatment
  Phase 2

SECONDARY OUTCOMES:
Number of participants with AEs | Up to approximately 2 years from end of treatment
  Phase 2
Number of participants with SAEs (as per CTCAE v5) | Up to approximately 2 years from end of treatment
  Phase 2
Number of participants with treatment-related adverse events (TRAEs) | Up to approximately 2 years from end of treatment
  Phase 2
Number of participants with AEs leading to discontinuation | Up to approximately 2 years from end of treatment
  Phase 2
Number of participants with AEs leading to death | Up to approximately 2 years from end of treatment
  Phase 2
Progression-free survival (PFS) by RECIST v1.1 per investigator assessment | Up to 4 years from randomization
  Phase 2
Duration of response (DOR) (PR or CR) by RECIST v1.1 per investigator assessment | Up to approximately 2 years from end of treatment
  Phase 2

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (71):
- United States (12):
  - Local Institution - 0117, New Haven, Connecticut
  - Local Institution - 0134, Washington D.C., District of Columbia
  - Local Institution - 0126, Orlando, Florida
  - Local Institution - 0124, Iowa City, Iowa
  - Local Institution - 0123, Baltimore, Maryland
  - Local Institution - 0094, St Louis, Missouri
  - Local Institution - 0096, Hauppauge, New York
  - Local Institution - 0127, Cleveland, Ohio
  - Local Institution - 0165, Charleston, South Carolina
  - Local Institution - 0114, Myrtle Beach, South Carolina
  - Local Institution - 0158, Salt Lake City, Utah
  - Local Institution - 0095, Seattle, Washington
- Argentina (2):
  - Local Institution - 0154, Buenos Aires
  - Local Institution - 0156, Buenos Aires
- Australia (4):
  - Local Institution - 0076, North Ryde, New South Wales
  - Local Institution - 0111, St Leonards, New South Wales
  - Local Institution - 0074, South Brisbane, Queensland
  - Local Institution - 0003, Malvern
- Local Institution - 0093, Brasília, Federal District, Brazil
- Canada (3):
  - Local Institution - 0007, Calgary, Alberta
  - Local Institution - 0109, Montreal, Quebec
  - Local Institution - 0009, Montreal, Quebec
- Chile (3):
  - Local Institution - 0105, Santiago, Santiago Metropolitan
  - Local Institution - 0005, Santiago, Santiago Metropolitan
  - Local Institution - 0163, Santiago
- Local Institution - 0052, Cali, Colombia
- Czechia (3):
  - Local Institution - 0147, Prague, Praha 5
  - Local Institution - 0149, Brno
  - Local Institution - 0150, Hradec Králové
- Finland (3):
  - Local Institution - 0044, Helsinki, Etelä-Suomen Lääni
  - Local Institution - 0029, Turku
  - Local Institution - 0060, Vantaa
- France (3):
  - Local Institution - 0083, Lille, Nord
  - Local Institution - 0080, Boredeaux
  - Local Institution - 0028, Villejuif
- Germany (4):
  - Local Institution - 0025, Jena, Thuringia
  - Local Institution - 0026, Hamburg
  - Local Institution - 0014, Herne
  - Local Institution - 0027, München
- Ireland (2):
  - Local Institution - 0059, Dublin
  - Local Institution - 0062, Dublin
- Italy (3):
  - Local Institution - 0139, Verona, Veneto
  - Local Institution - 0073, Milan
  - Local Institution - 0087, Napoli Campania
- Japan (3):
  - Local Institution - 0097, Koto-ku, Tokyo
  - Local Institution - 0078, Toyoma, Toyama
  - Local Institution - 0172, Fukuoka
- Mexico (6):
  - Local Institution - 0046, Monterrey, Nuevo León
  - Local Institution - 0048, Oaxaca City
  - Local Institution - 0122, Puebla City
  - Local Institution - 0049, Tlalpan
  - Local Institution - 0108, Tlalpan
  - Local Institution - 0118, Tlalpan
- Romania (4):
  - Local Institution - 0103, Cluj-Napoca
  - Local Institution - 0161, Craiova
  - Local Institution - 0100, Iași
  - Local Institution - 0101, Sibiu
- South Korea (3):
  - Local Institution - 0112, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0017, Seoul, Seoul-teukbyeolsi
  - Local Institution - 0167, Seoul
- Spain (3):
  - Local Institution - 0013, Madrid
  - Local Institution - 0091, Madrid
  - Local Institution - 0043, Seville
- Switzerland (3):
  - Local Institution - 0054, Chur
  - Local Institution - 0055, Sankt Gallen
  - Local Institution - 0056, Zurich
- United Kingdom (5):
  - Local Institution - 0057, Cardiff
  - Local Institution - 0019, London
  - Local Institution - 0063, London
  - Local Institution - 0020, Manchester
  - Local Institution - 0171, Sulton, Surrey

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07293351.html